CLINICAL TRIAL: NCT03156140
Title: Four Types of Pulse Oximeters Accurately Detect Hypoxia During Low Perfusion and Motion
Brief Title: Pulse Oximeter Motion Study
Acronym: Motion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Jennifer Lucero, Assistant Professor of Clinical Anesthesia, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pulse Motion
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia | interventions — Motion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- motion (Experimental): Right hand performs three different motion types
  Interventions: Other: Motion

INTERVENTIONS:
Other: Motion — Volunteer has motion on right hand while with continuous pulse oximetry during three oxygenation plateaus

SUMMARY:
Evaluate the performance of 4 pulse oximeters in 10 healthy adult volunteers with three motions compared to non-motion control at three arterial oxygen saturation target plateaus.

DETAILED DESCRIPTION:
Evaluate the performance of 4 pulse oximeters (Masimo Radical-7, Nihon-Koden OxyPal Neo, Nellcor N-600, and Philips Intellivue MP5) in 10 healthy adult volunteers. Three motions will be evaluated: tapping, pseudorandom, and volunteer-generated rubbing, adjusted to produce photoplethsmogram disturbance similar to arterial pulsation amplitude. During motion, inspired gases will be adjusted to achieve stable target plateaus of arterial oxygen saturation (SaO2) at 75%, 88%, and 100%. Pulse oximeter readings (SpO2) will be compared with SaO2 from simultaneous arterial blood samples

ELIGIBILITY:
Inclusion Criteria: healthy adult English speaking -

Exclusion Criteria: pediatric, cardiac or pulmonary condition. non-english speaking

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Pulse oximetry reading | immediate

SECONDARY OUTCOMES:
Arterial Blood gas | immediate

IPD SHARING:
Plan to Share IPD: No